CLINICAL TRIAL: NCT06845774
Title: Optimizing Low Threshold TelePrEP Care in Syringe Service Programs for People Who Inject Drugs in Appalachia
Brief Title: The PROTECT (PrEP Optimization Through Telehealth Care and Treatment) Trial
Acronym: PROTECT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hilary L Surratt, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Hilary L Surratt, PhD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90392; R34DA060087-01 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): One session standard of care (SOC) PrEP education (an in-use PrEP intervention based on CDC guidelines) with active referral to a local PrEP provider.
  Interventions: Behavioral: CDC PrEP with active referral
- Integrated Telehealth Care (Experimental): A multi-session PrEP education and intervention session that provides tailored PrEP education onsite combined with point-of-care PrEP testing and telehealth access to a PrEP provider.
  Interventions: Behavioral: TelePrEP

INTERVENTIONS:
Behavioral: CDC PrEP with active referral — The single session SOC utilizes structured risk assessments and educational materials recommended by the CDC, based on the CDC PrEP 101 information, and delivered one-on-one by trained study staff in about 15 minutes. This will be followed by active referral to a local provider; local providers have been identified to receive study referrals in each community. This session will occur the same day or within one week of study enrollment.
  Arms: Standard of Care
Behavioral: TelePrEP — The TelePrEP intervention includes an initial one-on-one in person intervention session with trained study staff that: 1) engages in provides basic education on PrEP care tailored for PWID; 2) encourages participation in a telehealth clinical evaluation for PrEP; and, 3) offers the opportunity to participate in point of care baseline testing for PrEP. At the conclusion of session 1, for those who express readiness to link with PrEP care, study staff will immediately facilitate access to the telehealth platform onsite. Four telehealth visits will be offered to access initial and follow-up clinical care for PrEP.
  Arms: Integrated Telehealth Care

SUMMARY:
The expansion of HIV pre-exposure prophylaxis (PrEP) care has been endorsed as a key strategy for reducing new HIV infections, however, PrEP trials among people who inject drugs (PWID) are rare and uptake of PrEP has been minimal, most notably in rural areas. Structural barriers to healthcare access, lack of providers, and inadequate infrastructure to deliver PrEP are challenges in many rural areas. In addition, PWID often have social determinant barriers to PrEP care. This study will integrate telehealth PrEP care within syringe services programs (SSPs), a venue already routinely accessed by PWID, to reduce structural barriers to evidence-based HIV prevention through co-located comprehensive PrEP services, and test this against a standard of care approach in a pilot randomized clinical trial. The primary objective is to examine preliminary efficacy and effect sizes of novel integrated telehealth care versus standard education and active referral on the primary outcome of PrEP initiation in HIV-negative participants who inject drugs.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* report at least one occasion of injection drug use in the past month
* report an indication for PrEP in the past six months consistent with CDC guidelines for PrEP care
* be a documented client of the county SSP at the time of study entry
* express willingness to participate in a multi-session intervention and follow-up

Exclusion Criteria:

* HIV-positive status
* current PrEP care.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
PrEP Initiation | 3 months post-baseline
  Number of participants initiating PrEP
PrEP Initiation | 6 months post-baseline
  Number of participants initiating PrEP

SECONDARY OUTCOMES:
PrEP Persistence | 3 months post-baseline
  Number of participants with PrEP prescription refill
PrEP Persistence | 6 months post-baseline
  Number of participants with PrEP prescription refill(s)
PrEP adherence | 3 months post-baseline
  Number of participants with tenofovir (TFV) detected in dried blood spot testing
PrEP adherence | 6 months post-baseline
  Number of participants with tenofovir (TFV) detected in dried blood spot testing

OTHER OUTCOMES:
Intervention Acceptability | 2 weeks post-baseline
  Level of Intervention Acceptability for the experimental arm; measured by 10 item Intervention Acceptability Questionnaire (IAQ) completed by participants post-intervention; range is 10-50, lower scores are higher satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Hilary L Surratt, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
REDCap de-identified survey data and clinical data from report forms will be preserved and shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study team will submit a de-identified and cleaned survey and clinical dataset to Dataverse at the completion of the project period, April 2027, or at publication of the primary outcomes paper, whichever is first.
Access Criteria: Data will be made available on the Harvard Dataverse, for which the University of Kentucky has an institutional account. The Harvard Dataverse Repository is a free data repository open to all researchers from any discipline, both inside and outside of the Harvard community, where investigators can share, archive, cite, access, and explore research data.